CLINICAL TRIAL: NCT07360964
Title: Clear Cell Chondrosarcoma in Italy: Insights Into Radiological, Clinical and pathologicaL Features, With Emphasis on Prognosis (CIRCLE)
Brief Title: Clear Cell Chondrosarcoma in Italy
Acronym: CIRCLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Azienda Ospedaliera Universitaria Pisana, Pisa (Unknown); Gaetano Pini CTO, Milano (Unknown); IRCCS Humanitas Research Hospital, Milano (Unknown); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); Ospedale "Morgagni - Pierantoni" di Forlì (Unknown); AOU Città della Salute e della Scienza Torino (Unknown); Azienda Consorziale Ospedaliero-Universitaria Policlinico di Bari (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIRCLE
Record Dates: First submitted 2026-01-08; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chondrosarcoma
Keywords: clear cell chondrosarcoma; prognosis
MeSH Terms: conditions — Chondrosarcoma; Chondrosarcoma, Clear Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients with a diagnosis of clear cell chondrosarcoma
  Interventions: Genetic: Molecular studies

INTERVENTIONS:
Genetic: Molecular studies — Molecolar studies to define possible prognostic parameters

SUMMARY:
Clear cell chondrosarcoma of bone is considered a low-grade malignant tumor in the last WHO classification of soft tissue and bone tumors; however, it is reported that recurrences and metastasis can occur. Considering the uncertain prognosis of this rare tumor, with some cases that historically seems to pursue a bad prognosis, we decided to collect all the Italian cases of clear cell condrosarcoma, in order to better understand its natural history and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with diagnosis of clear cell chondrosarcoma and chondrosarcoma with a clear cell component treated from 01 Jan 1982 to 31 Dec 2023
* Information available (date of primary tumor diagnosis, local treatments, systemic treatment, response to systemic treatment, date of progression) and date and status at last follow-up
* Imaging studies available for revision
* Histological slides available for revision

Exclusion Criteria:

* - Diagnosis different from clear cell chondrosarcoma or chondrosarcoma with a clear cell component;
* Absence of radiological and/or clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Prognostic accuracy | At baseline
  Ability of the model to predict overall survival, measured by AUC/C-index

CONTACTS AND LOCATIONS:
Locations (1):
- IRCC Rizzoli Orthopedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided